CLINICAL TRIAL: NCT00264095
Title: Blood Management Observation in Oncology Surgical Treatment (BOOST)
Brief Title: An Observational Study of Blood Management Techniques in Oncology Surgical Treatment
Status: Completed | Type: Observational
Sponsor: Janssen-Cilag B.V. (Industry)
Responsible Party: Sponsor
Other Study IDs: CR003460; EPOSUR4001
Record Dates: First submitted 2005-12-09; First posted 2005-12-12 (Estimated); Last update posted 2014-04-28 (Estimated); Status verified 2014-04

CONDITIONS: Anemia; Blood Loss, Surgical; Neoplasms
Keywords: Anemia; Blood loss; Transfusion; Blood transfusion; Erythropoietin; Surgery; Surgical blood loss; Tumor; Cancer; Surgical resection; Tumor resection
MeSH Terms: conditions — Anemia; Blood Loss, Surgical; Neoplasms; Hemorrhage

STUDY DESIGN:
Time Perspective: Cross-Sectional

GROUPS / COHORTS (1):
- 001
  Interventions: Procedure: Oncological surgery

INTERVENTIONS:
Procedure: Oncological surgery — surgery is primary observed intervention and blood loss is between 500-3000 ml

SUMMARY:
The purpose of this study is to observe the methods used to manage blood loss in surgical procedures to remove tumors from patients with cancer and to determine if there is a relationship with the need for blood transfusions.

DETAILED DESCRIPTION:
Considerable blood loss typically accompanies surgical procedures to remove malignant tumors. Blood transfusions, the best method of compensating for blood loss during surgery, have associated medical risks including infection transmission and allergic reaction, in addition to using significant amounts of red blood cells, which are often in short supply. Options exist to manage blood loss before surgery, including a procedure where a patient's own blood is stored in advance to be given if needed during surgery, and drug intervention, where a drug is given before surgery to help increase red blood cell production, thereby maintaining hemoglobin and oxygen levels in the body during surgery. This is a multi-center observational study to collect information regarding the methods used to manage blood loss in patients undergoing surgical removal of malignant tumors in the Netherlands. Information will be collected by study center and by patient over the course of approximately 18 months. For study center information, each observation period will last 2 months and there will be at least a 2-month interval between each observation period. For patient information there is one continuous observation period. General information regarding the frequency of use of different blood-saving techniques for the various types of operations performed will be collected from each of the centers participating in the study. Data obtained at the onset of the study will be compared to follow-up data gathered throughout the additional reporting periods and trends or changes in frequency of use of blood-saving techniques will be noted. The following information will be collected: medical history, tumor stage, type/site of operation, anticipated vs. actual blood loss during surgery, most recent hemoglobin and hematocrit values prior to the operation, blood-saving techniques used and the number of units and types of blood transfusions up to 24 hours after the operation. Information will be obtained from patients' medical records. No medication will be supplied by the study Sponsor and no specific procedures will be required for the study. Each patient's surgeon and anesthesiologist will be responsible for all decisions regarding his/her care and treatment during the operation. Information may be collected a maximum of one time from each patient during this study and there will be no follow-up information collected from individual patients. Since the study involves only the collection of information, no treatment will be required by the Sponsor and no medication will be supplied by the Sponsor.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a malignant tumor for which surgery is the first treatment
* Having an expected blood loss of at least 500 ml (100 teaspoons), and not more than 3000 ml (600 teaspoons)

Exclusion Criteria:

* Patients with a malignant tumor for which surgery is not the first treatment (i.e. have received chemotherapy first)
* Inability to speak, read and write Dutch

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a malignant tumour for which surgery is the primary treatment and a minimal blood loss of 500 ml. and a maximum blood loss of 3000 ml. is expected.
Sampling Method: Non-Probability Sample
Enrollment: 488 (Actual)
Dates: Start 2004-07; Primary Completion 2006-02 (Actual); Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
Patients' medical history; tumor stage; type/site of operation; anticipated vs. actual blood loss; hemoglobin/hematocrit values prior to surgery, blood-saving techniques used; number of units and types of blood transfusions up to 24 hours after surgery | 24 hours after surgery

SECONDARY OUTCOMES:
Frequency of use of different blood-saving techniques for the various types of operations performed from each of the centers participating in the study | within 24 hours after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag B.V. Clinical Trial, Study Director — Janssen-Cilag B.V.
Locations (11):
- Netherlands (11):
  - Alkmaar
  - Amersfoort
  - Apeldoorn
  - Deventer
  - Dordrecht
  - Drachten
  - Nieuwegein
  - Nijmegen
  - Roosendaal
  - Sneek
  - Zwolle